CLINICAL TRIAL: NCT01071317
Title: A Random Controlled Trial a Comprehensive Migraine Intervention at the Time of Discharge From the Emergency Department After Treatment for Acute Migraine
Brief Title: Trial of Comprehensive Migraine Intervention
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Benjamin W. Friedman, MD, Associate professor, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 09-08-248
Record Dates: First submitted 2010-02-17; First posted 2010-02-19 (Estimated); Results first posted 2018-07-26 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Naproxen; Sumatriptan

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Comprehensive care (Experimental): Reinforcement of diagnosis, education, medications, and referral
  Interventions: Drug: Naproxen; Drug: Sumatriptan; Behavioral: Migraine education; Behavioral: Reenforcement of diagnosis
- Typical care (Active Comparator): Usual care
  Interventions: Other: Typical care

INTERVENTIONS:
Drug: Naproxen — Naproxen 500mg PO bid prn headache
  Arms: Comprehensive care
Drug: Sumatriptan — 100mg po q day prn headache
  Arms: Comprehensive care
Behavioral: Migraine education — Educational program available through NIH/ national library of medicine/ X-plain
  Arms: Comprehensive care
Behavioral: Reenforcement of diagnosis — Patient advised has migraine headache and how the headache meets migraine criteria
  Arms: Comprehensive care
Other: Typical care — Care to be determined by attending physician
  Arms: Typical care

SUMMARY:
Despite the fact that more than 10% of Americans suffer from migraine, this headache disorder is often not diagnosed and not appropriately treated. The goal of this proposal is to determine whether a migraine protocol designed for use in an emergency room can be used to deliver the headache care that many migraine patients never receive. This is a randomized trial. Consecutive inadequately treated migraine patients will be randomized to TYPICAL care or to COMPREHENSIVE care. Those patients in the comprehensive care arm will receive the following intervention: 1) reinforcement of diagnosis, 2) an adaptable online educational intervention, reading material, and headache diaries, 3) two migraine specific medications and 4) expedited referral to a headache specialist, if needed. Patients in the typical care arm will receive whatever intervention the emergency physician feels is most appropriate. Headache surveys will be used toll if the protocol improves migraine-related pain and functional disability one month after the ER visit.

ELIGIBILITY:
Inclusion Criteria:

* Migraine,
* Baseline migraine related disability of mild or worse,
* No current or past triptan use,
* Not satisfied with current headache care.

Exclusion Criteria:

* Allergy or contraindication to study medications,
* Daily or near daily analgesic medication use.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Comprehensive Care: Reinforcement of diagnosis, education, medications, and referral
  Naproxen: Naproxen 500mg PO bid prn headache
  Sumatriptan: 100mg po q day prn headache
  Migraine education: Educational program available through NIH/ national library of medicine/ X-plain
  Reenforcement of diagnosis: Patient told he/s he has migraine headache and how the headache meets migraine criteria
Period: Overall Study
Arm/Group | Comprehensive Care | Typical Care
Started | 25 | 25
Completed | 23 | 23
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Population: Patients who enrolled and were randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Comprehensive Care | Typical Care | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (9) | 35 (9) | 34 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 20 | 43
  Male | 2 | 5 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50
Pre-existing migraine-related functional impairment as measured by the MIDAS scale [Median (Inter-Quartile Range); unit: units on a scale] — The Migraine Disability Assessment (MIDAS) Test is a brief, self-administered questionnaire designed to quantify headache-related disability over a 3 month period. It is a 5-question instrument used to determine the severity of the underlying migraine disorder. Each question is scored from 0 to 90; the total minimum and total maximum scores are 0 and 450 respectively. A total score of 0 indicates no impairment. A total score greater than 20 indicates severe migraine related functional impairment.
  units on a scale | 10 [7 to 18] | 13 [9 to 31] | 12 [9 to 25]

OUTCOME MEASURES:

1. Primary Outcome: Migraine Functional Impairment as Measured by Score on the Headache Impact Test 6 (HIT6) Scale
Description: This is a standardized instrument commonly used in migraine research. Participants answer 6 Likert questions about the impact of migraine on their daily life. A score of 36, the lowest possible score, indicates minimal functional impairment. A score of 78, the highest possible score, indicates substantial functional impairment
Time Frame: 1 month after study enrollment
Population: 2 patients in each group were lost-to-followup
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Comprehensive Care | Typical Care
Number analyzed (Participants) | 23 | 23
units on a scale | 59 [53 to 65] | 56 [51 to 62]

2. Secondary Outcome: Number of Participants Who Report Satisfaction With Treatment, as Measured by a Three Item Likert Scale
Description: Participants could report that they were completely satisfied, mostly satisfied or unsatisfied. Reported here are the number who were unsatisfied.
Time Frame: 1 month after study enrollment
Population: 2 patients in each group were lost to followup. One patient in the Typical Care group did not answer the question
Measure: Count of Participants; unit: Participants
Arm/Group | Comprehensive Care | Typical Care
Number analyzed (Participants) | 23 | 22
Participants | 4 | 4

3. Secondary Outcome: Number of Participants Who Report They Are Comfortable With Disease Management, as Measured by a Three-item Likert Scale
Description: Participants were asked to describe themselves as very comfortable, somewhat comfortable, or uncomfortable. Reported here are those who were very comfortable
Time Frame: 1 month after study enrollment
Population: Two patients in each arm were lost-to-follow-up. One patient in Typical Care did not answer this question.
Measure: Count of Participants; unit: Participants
Arm/Group | Comprehensive Care | Typical Care
Number analyzed (Participants) | 23 | 22
Participants | 10 | 6

4. Secondary Outcome: Number of Participants Who Returned to the Emergency Department for Management of Headache
Description: We report the number of patient who returned to the emergency department for management of headache
Time Frame: 1 month after study enrollment
Population: Two patients in each arm were lost to followup.
Measure: Count of Participants; unit: Participants
Arm/Group | Comprehensive Care | Typical Care
Number analyzed (Participants) | 23 | 23
Participants | 1 | 3

ADVERSE EVENTS:
Groups:
- Comprehensive Care: Reinforcement of diagnosis, education, medications, and referral
  Naproxen: Naproxen 500mg PO bid prn headache
  Sumatriptan: 100mg po q day prn headache
  Migraine education: Educational program available through HIH/ national library of medicine/ X-plain
  Reenforcement of diagnosis: Patient told he/s he has migraine headache and how the headache meets migraine criteria
Arm/Group | Comprehensive Care | Typical Care
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes